CLINICAL TRIAL: NCT03604705
Title: An Open-Label Study to Evaluate the Efficacy and Safety of APX001 in Non Neutropenic Patients With Candidemia, With or Without Invasive Candidiasis, Inclusive of Patients With Suspected Resistance to Standard of Care Antifungal Treatment
Brief Title: An Efficacy and Safety Study of APX001 in Non-Neutropenic Patients With Candidemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APX001-201; C4791009 (Other: Alias Study Number)
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Results first posted 2021-08-05 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Candidemia
MeSH Terms: conditions — Candidemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APX001 Treatment (Experimental)
  Interventions: Drug: APX001

INTERVENTIONS:
Drug: APX001 — APX001

SUMMARY:
This is a multicenter, open-label, non-comparative, single-arm study to evaluate the efficacy and safety of APX001 for the first-line treatment for candidemia including suspected or confirmed antifungal-resistant candidemia in non-neutropenic patients 18 yeas of age and older.

Suspicion of antifungal-resistant candidemia is sufficient (documented resistance is not required for enrollment). The Study Drug Treatment Period of APX001 will be a maximum of 14 days. After completion of 14 days study drug therapy, if further antifungal treatment is indicated to complete treatment of candidemia in accordance with standard practice guidelines, fluconazole (unless susceptibility results warrant alternative antifungal therapy) may commence for up to a further 7 days. There will be a Follow up Period of 4 weeks (+4 days) after EOT. The total duration of participation in the study is up to approximately 7.5 weeks.

This study will be conducted at approximately 20 sites in the United States and globally.

ELIGIBILITY:
Key Inclusion Criteria:

* Provision of written consent
* Adults ages 18 and above male or female
* New diagnosis of candidemia
* Able to have pre-existing intravascular catheters removed and replaced (as necessary)

Key Exclusion Criteria:

* neutropenia
* deep-seated Candida-related infections
* hepatosplenic candidiasis
* received more than 2 days of prior systemic antifungal treatment for current candidemia episode
* severe hepatic impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Engelhardt, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (29):
- United States (9):
  - University of Alabama at Birmingham School of Medicine, Birmingham, Alabama
  - University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - University of California, Davis, Davis, California
  - University of California-Davis Medical Center, Sacramento, California
  - Augusta University (Georgia Regents University), Augusta, Georgia
  - University of Chicago, Chicago, Illinois
  - Washington University, St Louis, Missouri
  - Duke University Hospital Medical Center, Durham, North Carolina
  - University of Texas- Health Science Center and Medical School at Houston, Houston, Texas
- Belgium (7):
  - Institut Jules Bordet,Service De Microbiologie, Brussels
  - Hopital Erasme, Brussels
  - Institut Jules Bordet, Brussels
  - Universite Libre de Bruxelles (ULB) - Hopital Erasme, Brussels
  - CHU de Charleroi - Hopital Civil Marie Curie, Lodelinsart
  - Mont-Godinne University Hospital, Yvoir
  - University Hospital Mont-Godinne, Yvoir
- Germany (3):
  - Klinik I fur Innere Medizin- Uniklinik Koln, Cologne
  - University Hospital Heidelberg, Heidelberg
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz - III. Medizinische Klinik Haematologie/Onkologie, Mainz
- Israel (6):
  - Infectious Diseases Unit, Rambam Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Infectious Diseases Unit, Tel Aviv
  - Sourasky Medical Center, Tel Aviv
  - Infectious Diseases Unit,Sheba Medical Center, Tel Litwinsky
  - Sheba Medical Center, Tel Litwinsky
- Spain (4):
  - Hospital Universitario Mutua de Terrassa, Terrassa, Barcelona
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital VLL D Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pappas PG, Vazquez JA, Oren I, Rahav G, Aoun M, Bulpa P, Ben-Ami R, Ferrer R, Mccarty T, Thompson GR, Schlamm H, Bien PA, Barbat SH, Wedel P, Oborska I, Tawadrous M, Hodges MR. Clinical safety and efficacy of novel antifungal, fosmanogepix, for the treatment of candidaemia: results from a Phase 2 trial. J Antimicrob Chemother. 2023 Oct 3;78(10):2471-2480. doi: 10.1093/jac/dkad256. PMID 37596890

RESULTS

PARTICIPANT FLOW:
Groups:
- APX001 Treatment: APX001: APX001 IV administration followed by APX001 oral tablet administration
Period: Overall Study
Arm/Group | APX001 Treatment
Started | 21
Completed | 20
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Treatment Period - MITT
Groups:
- Treatment Period - MITT: Evaluation of APX001 for the first-line treatment for candidemia, including suspected or confirmed antifungal-resistant candidemia, in non-neutropenic patients ≥ 18 years of age who had at least 1 positive blood culture within the 96 hours prior to starting study drug. Modified Intent-to-Treat (MITT) Population. The MITT Population contained 20 (95.2%) patients.
Arm/Group | Treatment Period - MITT
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 7
  United States | 3
  Israel | 9
  Spain | 1

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success at End of Study Treatment (EOST) as Determined by the Data Review Committee (DRC)
Description: Treatment Success is defined as meeting all of the following criteria:
  Two consecutive blood cultures negative for Candida spp. Alive at EOST No concomitant use of any other systemic antifungal therapies through end of study treatment
Time Frame: One to forty-two days
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Period - MITT: Treatment Success was defined as meeting all of the following criteria: 1) 2 consecutive blood cultures were negative for Candida spp.; 2) Alive at EOST; and 3) No concomitant use of any other systemic antifungal therapies through EOST. Treatment Failure is defined as any case that does not meet the criteria for Treatment Success.
Arm/Group | Treatment Period - MITT
Number analyzed (Participants) | 20
Participants | 16

2. Secondary Outcome: Time to First Negative Blood Culture
Description: Time to first negative blood culture was defined as the number of days from first dose date of study drug to the date of first post-Baseline negative blood culture + 1. Patients without a negative blood culture at post-Baseline visits were censored at the last assessment date.
Time Frame: One to forty-nine days
Measure: Mean (Standard Deviation); unit: Days
Groups:
- MITT Population: MITT = Modified Intent-to-Treat population
Arm/Group | MITT Population
Number analyzed (Participants) | 20
Days | 2.4 (1.13)

3. Secondary Outcome: Percentage of Patients With Mycological Outcomes at End of Study Treatment (EOST), End of Treatment (EOT), and 2 and 4 Weeks After End of Treatment (EOT)
Time Frame: End of study treatment (EOST), end of treatment (EOT), and 2 and 4 weeks after end of treatment (EOT)
Measure: Count of Participants; unit: Participants
Groups:
- EOST (End of Study Drug Treatment); EOT (End of Antifungal Treatment): Eradication
- Follow-up 2 Weeks After EOT; Follow-up 4 Weeks After EOT: Recurrence
Arm/Group | EOST (End of Study Drug Treatment) | EOT (End of Antifungal Treatment) | Follow-up 2 Weeks After EOT | Follow-up 4 Weeks After EOT
Number analyzed (Participants) | 20 | 20 | 20 | 20
Participants | 16 | 15 | 1 | 0

4. Secondary Outcome: Percentage of Patients With Treatment Success at End of Treatment (EOT), and 2 and 4 Weeks After End of Treatment (EOT)
Time Frame: 2 and 4 weeks after end of treatment (EOT)
Measure: Number; unit: percentage of participants
Groups:
- Treatment Success 2 Weeks After EOT; Treatment Success 4 Weeks After EOT: Treatment Success determined by the DRC by visit for the MITT Population.
Arm/Group | Treatment Success 2 Weeks After EOT | Treatment Success 4 Weeks After EOT
Number analyzed (Participants) | 20 | 20
percentage of participants | 60.0 | 55.0

5. Secondary Outcome: Overall Survival at Study Day 30
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | MITT Population
Number analyzed (Participants) | 20
Participants | 17

6. Secondary Outcome: Number of Patients With Treatment Emergent Adverse Events (TEAEs)
Time Frame: One to forty-nine days
Measure: Count of Participants; unit: Participants
Groups:
- Safety Population: Twenty-one patients were dosed with APX001 and composed the ITT/Safety Population.
Arm/Group | Safety Population
Number analyzed (Participants) | 21
Participants | 20

ADVERSE EVENTS:
Time Frame: One to forty-nine days
Arm/Group | Safety Population
All-Cause Mortality (participants affected / at risk) | 5/21
Serious Adverse Events (participants affected / at risk) | 9/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=21)
Septic shock (Infections and infestations) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1)
Enterobacter sepsis (Infections and infestations) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Stenotrophomonas sepsis (Infections and infestations) | 1 (1)
Systemic candida (Infections and infestations) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Euthanasia (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=21)
Bacteraemia (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Oedema peripheral (General disorders) | 3 (3)
Pyrexia (General disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT03604705/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT03604705/SAP_001.pdf